CLINICAL TRIAL: NCT06859372
Title: Nurturing Care Family Navigator: Establishing Practices for Navigating Maternal-Child Food Insecurity
Brief Title: Nurturing Care Family Navigator
Acronym: NCFN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Gabriela Buccini, Assistant Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: UNLV-2024-424; U01HD115256 (NIH); U01OD033239 (NIH)
Record Dates: First submitted 2025-01-16; First posted 2025-03-05 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Food Insecurity Among Children; Food Insecurity in Post Partum Women; Care Coordination in Primary Care; Preventive Care / Anticipatory Guidance; Retention in Care
Keywords: Maternal-Child Health; Food Insecurity; Navigation; Postpartum; Pediatrics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Non-Navigation Cohort (No Intervention): Participants in the control group will receive an educational workbook with messages across the four pillars of food insecurity (standard of care). Non-navigation will be provided.
- Experimental: Navigation Group (Experimental): Participants who are randomized into the NCFN program will be assigned to a navigator. The NCFN will deliver the behavioral health navigation intervention consisted an educational workbook (standard of care) plus a total of 15 sessions tailored to the participant needs. The NCFN will offer support and referral to community resources (e.g., food, transportation, housing, healthcare-related). The navigator will provide intense weekly educational support and linkage to resources during the initial three months of the program and additional monthly follow up sessions during the last three months of the program.
  Interventions: Behavioral: Nurturing Care Family Navigator

INTERVENTIONS:
Behavioral: Nurturing Care Family Navigator — The Nurturing Care Family Navigator (NCFN) is a comprehensive barrier-focused and long-term family-centered intervention that will offer screenings for food insecurity, referrals to community resources, and follow-up with families experiencing very low or low food security in the past 12 months. The goal of the NCFN is to increase knowledge (cognitive factors) and self-efficacy (behavioral factors) to navigate barriers across the four pillars of food insecurity by securing enrollment and sustaining engagement with a set of community nurturing care services (environmental factors) to improve levels of food security, and ultimately maternal-child health and nutrition outcomes of low-income families during the postpartum phase.
  Arms: Experimental: Navigation Group

SUMMARY:
The goal of this pilot randomized controlled trial is to determine whether a 6-month behavioral health intervention with a Nurturing Care Family Navigator (NCFN) improves levels of food security among postpartum low-income Medicaid or uninsured women identified as having very low or low food security in the past 12 months. We hypothesize that a behavioral health intervention applying a multisectoral nurturing care navigation approach facilitating access to health, nutrition, early learning, responsive care, and security and safety resources is likely to decrease levels of maternal-child food insecurity. The main question it aims to answer is:

* Does the behavioral health intervention with a Nurturing Care Family Navigator (NCFN) improves levels of food security? Outcome 1: Improve levels of food security
* Does the behavioral health intervention with a Nurturing Care Family Navigator (NCFN) increase knowledge to navigate barriers across the four pillars of food insecurity? Outcome 2: Increase knowledge across the four pillars of food insecurity
* Does the behavioral health intervention with a Nurturing Care Family Navigator (NCFN) increase self-efficacy to secure and sustain enrollment with community nurturing care services? Outcome 3: Increase self-efficacy to secure and sustain enrollment with community nurturing care services

Researchers will compare levels of food security among those receiving a navigation behavioral health intervention (consisted of 1:1 tailored navigation session and an educational workbook) compared to those receiving an educational workbook with messages across the four pillars of food insecurity (standard of care).

Participants will:

* Engage in intense weekly navigation 1:1 tailored session for 3 months
* Engage in follow up monthly navigation 1:1 tailored session for 3 months
* Participate in evaluation calls with a research assistant at enrollment, 3, 6, 12 months

DETAILED DESCRIPTION:
The Nurturing Care Family Navigator (NCFN) is a social behavioral health intervention inspired by the Nurturing Care Framework which provides an evidence-based roadmap across and within five components (i.e., health, nutrition, early learning, security and safety, and responsive caregiving) to transform child rights into equitable actions to address threats and promote optimal early childhood development. We hypothesize that applying a multisectoral nurturing care navigation approach facilitating access to health, nutrition, early learning, responsive care, and security and safety community resources is likely to decrease levels of maternal-child food insecurity.

The NCFN is the navigation program under investigation. NCFN is a comprehensive barrier-focused and long-term family-centered intervention that will offer screenings for food insecurity, referrals to community resources, and follow-up with families experiencing very low or low food security in the past 12 months assessed using the 8-item Abbreviated Child and Adult Food Security Scale (ACAFSS). The NCFN program is grounded in the Social Cognitive Theory (SCT) aiming to support families in overcoming barriers within and across the four pillars of food security (i.e., food availability, access to food, utilization, and stability). The goal of the NCFN is to increase knowledge (cognitive factors) and self-efficacy (behavioral factors) to navigate barriers across the four pillars of food insecurity by securing enrollment and sustaining engagement with a set of community nurturing care services (environmental factors) to improve levels of food security, and ultimately maternal-child health and nutrition outcomes of low-income families during the postpartum phase.

The target population for the randomized controlled trial will consist of (1) low-income Medicaid or uninsured families with an infant one week postpartum attending the well child visit at a Pediatric clinic through UNLV Health; (2) identified as having very low or low food security in the past 12 months; and (3) residing in one of the zip codes within Clark County, Nevada. The intervention group will receive the NCFN program that will support families through 15 one-on-one sessions over 6 months after enrollment (a total of 15 sessions with 12 sessions in the first 3 months and 3 sessions in the last 3 months) and one year of follow up evaluation with a research assistant. The control group will receive an education workbook package and one year of follow up evaluation with a research assistant. Participants will undergo surveys at enrollment, three, six, and 12 months after enrollment (i.e., baseline, T2, T3, T4). Additionally, the research team will conduct interviews with navigators as well as clinical and non-clinical providers.

ELIGIBILITY:
Inclusion Criteria:

* Individuals postpartum low-income, Medicaid publicly funded or uninsured
* Individuals 18 years or older
* Individuals with infants up to two weeks postpartum
* Ability to speak and read English or Spanish
* Established patient at the UNLV Pediatric (at least one well-child visit)
* Lives in one of the zip codes within Clark County, Nevada, United States

Exclusion Criteria:

* Intent to transfer care to an institution other than UNLV Pediatric
* Infants who receive at birth any of the following diagnoses: Down syndrome, cleft lip and/or palate, congenital heart disease, neurological conditions, and cardiac problems.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Intense Navigation Completion | T2 (3 months)
  Number of NCFN sessions completed (range 0-12). Engage in a total of 12 one-on-one session over three-months. Navigation interruptions/stoppages were considered incomplete intervention. A 90% navigation completion rate was chosen a priori to indicate a promising intervention.
Follow Up Navigation Completion | T3 (6 months)
  Engage in a total of 3 follow up session over three-months after the end of the intense intervention (range 0-3). Number of follow-up sessions completed. A 90% navigation completion rate was chosen a priori to indicate a promising intervention.
Navigation Completion | T3 (6 months)
  Engage in a total of 15 one-on-one session over six-months. Navigation interruptions/stoppages were considered incomplete intervention. A 90% navigation completion rate was chosen a priori to indicate a promising intervention.
Food Security Status Baseline | Baseline
  Food security status will be determined by the sum of affirmative responses to the 8-item Abbreviated Child and Adult Food Security Scale (ACAFSS) in the past 12 months. ACAFSS scores range from 0 to 8. Higher scores represent greater food insecurity: 0-1 means the household is food secure; 2-4 means the household is low food security; 5-8 means the household is very low food security.
Food Security Status Point 1 | Baseline and T2 (3 months)
  Food security status will be determined by the sum of affirmative responses to the 8-item Abbreviated Child and Adult Food Security Scale (ACAFSS) in the past 30 days. ACAFSS scores range from 0 to 8. Higher scores represent greater food insecurity: 0-1 means the household is food secure; 2-4 means the household is low food security; 5-8 means the household is very low food security. Changes in scores and food security status will be examined between Baseline and T2 (3 months).
Food Security Status Point 2 | Baseline and T3 (6 months)
  The unabbreviated scale used to measure the participants' food security status is the Abbreviated Child and Adult Food Security Scale (ACAFSS), validated for 12 months and 30 days in the United States population. ACAFSS scores range from 0 to 8. Higher scores represent greater food insecurity: 0-1 means the household is food secure; 2-4 means the household is low food security; 5-8 means the household is very low food security. Changes in scores and food security status will be examined between Baseline and T3 (6 months)
Food Security Status Point 3 | Baseline and T4 (12 months)
  The unabbreviated scale used to measure the participants' food security status is the Abbreviated Child and Adult Food Security Scale (ACAFSS), validated for 12 months and 30 days in the United States population. ACAFSS scores range from 0 to 8. Higher scores represent greater food insecurity: 0-1 means the household is food secure; 2-4 means the household is low food security; 5-8 means the household is very low food security.Changes in scores and food security status will be examined between Baseline and T4 (12 months)

SECONDARY OUTCOMES:
Patient reported Perceived Barriers to Food Security | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  The Barriers Needs Assessment Form is a non-validated questionnaire created by the research team to assess perceived barriers to food security such as personal, food, transportation, healthcare, infant, housing, and resource concerns. By systematically identifying perceived barriers, the intervention can implement targeted strategies to address them, such as connecting participants with community resources.The questionnaire was designed with yes/no questions and range from 0 to 52 perceived barriers. Higher scores represent greater perceived barriers. The questionnaire will assess perceived barriers in the intervention and control groups at each time point: baseline T2 (3 months), T3 (6 months), and T4 (12 months).The assessment of perceived barriers will be used to document changes across different time points.
Patient-reported Self-Efficacy for Food Security Scale | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  The Self-Efficacy for Food Security Scale is a validated questionnaire designed to assess an individual's confidence in their ability to access and maintain a sufficient and nutritious food supply despite potential challenges. Responses range from 1-4 and they are recorded on a Likert scale ranging from "not at all confident" to "very confident", allowing for an assessment of self-efficacy levels. Higher scares indicate greater self-efficacy: 3-4 indicates high self-efficacy and 1-3 indicates low self-efficacy. The questionnaire will assess both the intervention and control groups at each time point: baseline T2 (3 months), T3 (6 months), and T4 (12 months).The assessment of self-efficacy will be used to document changes across different time points.
Patient-reported Perceived Agency ("Seeking" Behavior) | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  Differences in "seeking" behavior assessed by the agency questionnarie at baseline, T2 (3 months), T3 (6 months), T4 (12 months).The perceived agency questionnaire was adapted by the research team. It consists of five questions, and each question is scored on a 3-point scale between 1 and 3. Total scores ranges from 5 to 15. Higher scores indicate greater agency/seeking behavior.
Patient-reported Maternal Diet Quality Index | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  Maternal diet quality reported through the validated Rapid Prime Diet Quality Score Screener (rPDQS).The RPDQS Screener is a brief dietary assessment tool designed to quickly evaluate diet quality based on key food groups associated with health outcomes. It consists of a short questionnaire of 13 questions assessing the consumption of beneficial and harmful food groups and one evaluation of alcohol consumption. The scoring system is a numeric scoring approach that allocates 0 to 4 points to consumption of each of the six food groups whose intake is encouraged (with a reverse scoring for the seven food groups to limit) based on the original frequency of consumption (range, 0-52; higher = healthier).
Patient-reported Breastfeeding Status | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  Total duration of exclusive or partial breastfeeding at enrollment, 3 months, 6 months, and 12 months
Patient-reported Infant Feeding | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  Infant feeding quality assessed through the World Health Organization Infant. This questionnaire allows to assess a set of indicators to assess infant and young child feeding.

OTHER OUTCOMES:
Patient-reported Postpartum Depression Screening using Edinburgh Postnatal Depression Scale (EPDS) | Baseline, T2 (3 months)
  The Edinburgh Postnatal Depression Scale (EPDS) is a validated to screen for symptoms of postpartum depression (PPD) in new mothers. The EPDS consists of 10 questions assessing emotional well-being over the past seven days. Each question is scored on a 4-point scale between 0 and 3, with total scores ranging from 0 to 30. Higher scores indicate a greater likelihood of depressive symptoms. The scale includes items related to sadness, anxiety, guilt, sleep disturbances, and thoughts of self-harm, making it effective in detecting both symptoms of depression and postpartum anxiety.
Patient-reported Postpartum Depression Symptoms using the Patient Health Questionnaire (PQH-9) | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  Participants will be screened for depression using the Patient Health Questionnaire (PQH-9). The PQH-9 relies on patients self-reporting nine items regarding their health in the past two weeks. Each question is scored from 0 (not at all) to 3 (nearly every day), with a total possible score of 27. A score of 10 or higher will be considered a positive screen for depression.
Patient-reported Anxiety Symptoms using the General Anxiety Disorder-7 (GAD-7) | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  Participant screened for anxiety using the General Anxiety Disorder-7 (GAD-7). The GAD-7 relies on patients self-reporting seven items regarding their health in the past two weeks. Each question is scored from 0, 1, 2, and 3 to the response categories, respectively, of "not at all," "several days," "more than half the days," and "nearly every day." 0 (not at all) to 3 (nearly every day). GAD-7 total score for the seven items ranges from 0 to 21. Higher scores indicates severity of anxiety symptoms: 0-4: minimal anxiety, 5-9: mild anxiety, 10-14: moderate anxiety, 15-21: severe anxiety.
Patient-reported Stress using the Postpartum Stressors Scale (PPSS) | Baseline
  Participant screened for stress using the Postpartum Stressor Measure. A 9-item scale that measures stress in three areas: baby care, well-being, and work problems. Each question is scored from 0 (not at all) to 4 (very stressful). The score ranges from 9-36. Higher scores reflect higher stress.
Patient-reported Perceived Discrimination using the Perceived Personal Discrimination in Interactions with Healthcare Providers | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  Perceived Personal Discrimination in Interactions with Healthcare Providers is a validated self-report questionnaire that measures patients' experiences of discrimination, such as being dismissed, treated with less respect, or receiving lower-quality care. The questionnaire assess seven questions using Likert-scale responses that range from "never" to "always" to gauge the frequency and intensity of discriminatory encounters. The range of possible scores would be 7-35, with a higher number indicating more perceived discrimination.
Patient-reported Social Support using Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  The "General Social Support: MSPSS" refers to the "Multidimensional Scale of Perceived Social Support" which is a 12-question self-report questionnaire where each question is rated on a 7-point Likert scale, meaning individuals choose a response ranging from "strongly disagree" to "strongly agree" to assess their perceived level of social support from family, friends, and significant others. Higher scores means higher perceived support:12 - 35 Low perceived support, 36-60 Medium perceived support; 61-84 High perceived support. Changes in social support category will be assessed at baseline, T2 (3 months), T3 (6 months), T4 (12 months).
Patient-reported Perceived Nutrition Environment | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  Changes in perceived nutrition environment will be assessed at baseline, T2 (3 months), T3 (6 months), T4 (12 months). Survey items were adapted from the validated Perceived Nutrition Environment Measures Survey (NEM-P). The research team selected 25 items to assess relevant constructs to the intervention: consumer nutrition environment, community nutrition environment, background characteristics, and food shopping behaviors. Higher scores means higher perceived nutrition environment.
Patient-reported Satisfaction with Navigator Interpersonal Relationship (PSN-I) | T2 (3 months)
  Navigated participants' experiences with navigation as assessed through the validated Patient Satisfaction with Interpersonal Relationship with Navigator (PSN-I) scale. The scale contains 9 items scored as a Likert scale with each item ranging from 1-4. Lower PSN-I total score indicates higher satisfaction.
Program data - Number of referrals | T2 (3 months), T3 (6 months), T4 (12 months)
  Program data will be used to quantify the number of referrals made, referrals connected (warm hand-off), and referrals enrolled.
Program data - Participation in community workshops | T2 (3 months), T3 (6 months), T4 (12 months)
  Program data will be used to quantify the number of workshops participants engaged throughout 12 months.
Program data - Number of Resources Enrolled | Baseline, T2 (3 months), T3 (6 months), T4 (12 months)
  Program data will be used to quantify the number of resources participant is enrolled. The difference in number of resources participant is enrolled from baseline to end of study. A non-validated questionnaire will be used to collect information on resources' enrollment. Resources will be classified in food-related resources enrolled, health-related resources enrolled, and other types of resources enrolled.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD and all IPD that underlie results will be made available in publications.
Supporting Information: Study Protocol, ICF